CLINICAL TRIAL: NCT07194512
Title: The Effect of Eight Weeks of High-Intensity Interval Training on Physical Performance in Young Taekwondo Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Ali Osman Kıvrak, Associate Professor, Selcuk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SelcukU--SBF-AEB-AOK-2025-001
Record Dates: First submitted 2025-09-07; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Hight Intensity Interval Training
Keywords: Agility; explosive power; Hight intensity interval training; Sport-specific test; taekwondo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Two groups (Other): "Experimental group" and "Control group"
  Interventions: Other: Taekwondo-Specific Agility Test (TSAT), Frequency Speed of Kick Test (FSKT), Frequency Speed of Kick Test (FSKT10s), Multiple Frequency Speed of Kick Test (FSKTmult), Kick Decrement Index (KDI)

INTERVENTIONS:
Other: Taekwondo-Specific Agility Test (TSAT), Frequency Speed of Kick Test (FSKT), Frequency Speed of Kick Test (FSKT10s), Multiple Frequency Speed of Kick Test (FSKTmult), Kick Decrement Index (KDI) — After pre-test measurements, the experimental group performed an eight-week high-intensity interval training (HIIT) program three times per week (Monday, Wednesday, Friday) alongside their regular taekwondo training. The control group continued with their regular taekwondo training only. After the eight-week intervention, post-tests were administered to both groups, and the results were recorded by the researchers.

SUMMARY:
The goal of this clinical trial is to determine the effects of an eight-week high-intensity interval training program on agility, frequency speeds of kick, vertical jump, and standing long jump performances in young taekwondo. The main question it aims to answer is: Our main hypothesis is that the 8 week high-intensity interval training program improve agility, frequency speeds of kick, vertical jump, and standing long jump performances of young taekwondo Researchers will compare the experimental group and control group to see if the training program improve the agility, frequency speeds of kick, vertical jump, and standing long jump performances.

Participants will perform the 8 week hight inntesity interval training.

ELIGIBILITY:
Twenty male taekwondo athletes aged 16 to 18 from Süer Sports Club in Ankara participated in the study.

Inclusion Criteria: When forming the groups, care was taken to ensure that none of the athletes were currently undergoing injury rehabilitation or had any recent injuries that could affect their performance. Additionally, all voluntary participants underwent health screening to verify their current health status.

Exclusion Criteria: Athletes with injuries or illnesses were not included in the study.

Ages: 16 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Taekwondo-Specific Agility Test (TSAT) | For 8 weeks from the start of the study
  As previously described, the test begins with the athlete in a guard position, with both feet positioned behind the starting/finishing line, and proceeds sequentially as follows:
  1. The athlete must move as quickly as possible into the center point while maintaining the guard position.
  2. The athlete must change direction, turn toward Partner 1, and perform a Palding kick with the left leg.
  3. The athlete must move toward Partner 2 and perform a Dollyo-Chagi kick with the right leg.
  4. The athlete must return to the center.
  5. The athlete must move forward in the guard position, and perform a Double Palding kick toward Partner 3.
  6. Finally, the athlete must return to the starting/finishing line while maintaining the guard position.
Frequency Speed of Kick Test (FSKT10s) | For 8 weeks from the start of the study
  To assess the best possible single FSKT score, athletes were subjected to the FSKT10s. In this test, athletes were instructed to perform as many mid-level kicks as possible within a 10-second period, with the total number of valid kicks recorded as the score. Following a five-minute rest, the protocol was repeated, and the best score from the two trials was recorded as the FSKT10s . According to the FSKT classification, athletes who performed 16 or fewer kicks were classified as "very poor," those with 17 kicks were categorized as "poor," 18-21 kicks as "average," 22-23 kicks as "good," and 24 or more kicks were classified as "excellent".
Multiple Frequency Speed of Kick Test (FSKTmult) | For 8 weeks from the start of the study
  To assess the athletes' FSKTmult scores, the FSKT test was conducted in five consecutive sets, with 10-second rest intervals between each set. Each set consisted of the maximum number of kicks the athletes could perform within 10 seconds, as previously described. At the end of the five sets, the total valid kicks performed by the athletes in each set (FSKT1, FSKT2, FSKT3, FSKT4, FSKT5) and the overall total (FSKT5x10s total) were recorded for analysis.
Kick Decrement Index (KDI) | For 8 weeks from the start of the study
  To indicate performance decrement in the FSKT5x10s test, the KDI (%) ratio was used. This ratio incorporates the number of kicks performed in each set and the potential maximum number of kicks, calculated using the equation provided below.
  KDI (%) = [1-(FSKT_1+FSKT_2+FSKT_3+FSKT_4+FSKT_5)/(Best FSKT x Number of Sets)] x 100
Vertical Jump Test | For 8 weeks from the start of the study
  The TKK 5406 jump meter was used to apply the vertical jump test. Prior to the test, athletes were allowed sufficient repetitions to familiarize themselves with the equipment. During the test, athletes were instructed to stand with both feet on the mat of the measurement device and jump as high as possible when the device's light signal was activated. Arm and leg swings were permitted during the jump. Care was taken to ensure that athletes landed on both feet simultaneously. The vertical jump distance for each athlete was recorded from the device's display after the jump. The test was repeated three times, with a 1-minute rest interval between attempts. The best jump from the three trials was recorded as the athlete's vertical jump performance.
Standing Long Jump Test | For 8 weeks from the start of the study
  Athletes were positioned with their toes just behind the starting line, feet at a normal width, and with their arms extended forward and knees bent in a pre-jump stance. They were instructed to jump as far as possible, using their arms for momentum, and both feet were to land simultaneously. The distance from the starting line to the athlete's heels was measured in centimeters and recorded. Athletes were given two attempts, and the best result was taken for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Osman Kıvrak, Associate Professor, Principal Investigator — Department of Coaching Education, Faculty of Sport Sciences, Selçuk University
Locations (1):
- Alaeddin Keykubat Yerleşkesi Akademi Mah. Yeni İstanbul Cad. Selçuklu, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided